CLINICAL TRIAL: NCT03791541
Title: A Study Evaluating the Use of Potential Predictors of Readmission in Hospitalized Medicine Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study results not meaningful. Students researchers graduated.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mathew Thambi, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0748
Record Dates: First submitted 2018-12-20; First posted 2019-01-02 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: The Focus is to Test a Survey Predicting Readmissions; Inpatient Internal Medicine Patients
Keywords: Readmissions; Survey

STUDY DESIGN:
Intervention Model Description: targeted, cost-effective interventions based on results of surveys and other factors studied will be applied to study arm to see if re-admissions can be prevented
Who Masked: Participant
Masking Description: Survey will be given to all participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Only surveys will be done and re admissions tracked. No additional interventions based on survey results will be done.
- Intervention (Experimental): Pharmacist Services
  Surveys plus increased outpatient pharmacist/pharmacy student services including but not limited to pre and post clinic visit phone calls, prescription counseling, and helping with adherence and compliance with medications. Increased services will be given based on survey results.
  Interventions: Behavioral: Pharmacist services

INTERVENTIONS:
Behavioral: Pharmacist services — Additional pharmacist/pharmacy student follow-ups, counseling, and other services
  Arms: Intervention

SUMMARY:
The primary objective of this study is the development and implementation of a survey administered to hospitalized patients on Internal Medicine that can be used in conjunction with previously validated predictive indices to identify patients at risk for readmission. The survey consists of previously validated as well as investigator developed survey instruments that will assess the following: health literacy, numeracy, medication adherence, self-efficacy, and tolerance. The predictive indices are the LACE, Charlson Comorbidity Index (included in LACE), and the Comorbidity Polypharmacy Score (CPS) which have been previously validated for risk of readmissions. The survey consists of both closed and open ended questions. A part of the survey will be administered by the study personnel while the rest is a questionnaire-based survey that will be completed by the subjects. Study personnel will be with the subjects in an open dialogue while subjects are completing the survey to answer any questions and identify questions that may be confusing or bias subjects. Approximately 30 days after hospital discharge, patients will be contacted via telephone to ask how many admissions and/or Emergency Department (ED) visits they have had since discharge. A correlation analysis will be done of the different aspects of the survey to determine whether there are redundancies. A regression analysis will be done to determine the predictive ability of the survey combined with predictive indices for readmission.

DETAILED DESCRIPTION:
Many patients are readmitted to the hospital shortly after discharge. Twenty percent of Medicare beneficiaries discharged were re-hospitalized within 30 days at a cost to Medicare estimated at $17.4 billion. This problem does not only affect the elderly. Medicaid enrollees aged 21-64 had 10.7% 30-day readmission rate. Identifying which patients are at highest risk is important for allocating resources to those high risk individuals.

Several studies have attempted to retrospectively identify medical conditions, medications, labs, and vitals associated with increased risk of readmission with different levels of success. Examples of these include the Charlson Comorbidity Index, LACE, and the Comorbidity Polypharmacy Score. Although not always developed for use in predicting readmissions, they have been subsequently associated with this.

While these indices examine objective data, it is thought that health beliefs, abilities, and behaviors can also affect the risk of readmissions. Health literacy in particular has been shown to be associated with 30 day readmissions after an acute myocardial infarction and in general medical patients. Low numeracy has been associated with increased risk of 30 day readmission in patients with acute heart failure.

Inpatient questionnaires are able to identify patients who are more likely than others to be readmitted. Additionally, objective qualities such as insurance status, comorbidities, and admissions within the past year are predictors of readmission. Due to the unique patient populations at different health systems, an institution-specific approach is necessary to analyze the specific factors contributing to readmission. Therefore, a survey will be used to gauge the most predictive factors of readmissions and ED visits, including objective and subjective sections. After further research and modification, the survey will potentially serve as a tool for clinicians to select the best approach to post-discharge care and follow-up.

This pilot will attempt to test a survey for predicting readmission through measurements of health literacy, numeracy, medication adherence, self-efficacy, and tolerance, and in conjunction with co-morbidity indices.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient on Internal Medicine service at UIH (University at Illinois Health Hospital)
* Adults > 18 years of age, fluency in English

Exclusion Criteria:

* Prisoners
* Active illicit substance abuse per admitting History & Physical note in EMR (Electronic Medical Record)
* Admitted for alcohol withdrawal or abuse
* Nursing home resident likely to be discharged back to a nursing home
* Unable to provide informed consent
* Unable to complete survey (e.g., dementia)
* Unable to communicate verbally (aphasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Number of readmissions after 1 month | 30 days post-discharge
  Number of readmissions after 30 days post-discharge

SECONDARY OUTCOMES:
Number of readmissions after 2 months | 60 days post-discharge
  Number of readmissions after 60 days post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mat Thambi, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No